CLINICAL TRIAL: NCT00146380
Title: A Phase II Open Label Clinical Trial of Maternal Zidovudine/Lamivudine and Either Nevirapine or Nelfinavir for Maximal Reduction of Mother-to-child HIV Transmission in Resource-limited Settings Among Breastfeeding Populations
Brief Title: A Study of Zidovudine/Lamivudine and Either Nevirapine or Nelfinavir for Reduction of Mother-to-child HIV Transmission During Breastfeeding
Acronym: KiBS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHSTP-3677; UR6/CCU018970
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: HIV Infections
Keywords: Prevention Mother-to-Child HIV transmission; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine; Lamivudine; Nelfinavir; Lactation; Postpartum Period

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Zidovudine/Lamivudine and either Nevirapine or Nelfinavir — Zidovudine 300mg po bid from 34 weeks gestation to 6 months postpartum Lamivudine 150mg po bid from 34 weeks gestation to 6 months postpartum AND EITHER Nevirapine 200mg po qd for 2 weeks as lead in then bid from 34 weeks gestation to 6 months postpartum OR Nelfinavir 1250mg po bid from 34 weeks gestation to 6 months postpartum
  ARVs continued for those that meet WHO treatment criteria
Behavioral: Breastfeeding for 6 months postpartum — Exclusive breastfeeding till five and one half months with rapid weaning over 2 weeks and cessation of breastfeeding at 6 months when ARVs are discontinued

SUMMARY:
The purpose of the study is to demonstrate that a regimen using highly active antiretroviral therapy (HAART) to maximally suppress maternal viral load in the late antenatal period and during the first six months of lactation is safe, effective and can be implemented in resource poor settings in order to reduce the risk of HIV transmission to the infant.

DETAILED DESCRIPTION:
Background: Approximately 800,000 HIV-infected infants are born each year, two thirds of them in sub-Saharan Africa. The rate of HIV transmission from mother to infant is estimated at 13-48% in the absence of antiretroviral treatment. Interventions currently available to prevent mother to child transmission in resource-limited settings among breastfeeding populations child HIV transmission during the breastfeeding period. Because safe alternatives to breastfeeding are not currently a viable option for many HIV-infected women in sub-Saharan Africa, it is important to identify interventions to decrease transmission to the infant during this period.

Objective: To demonstrate that a regimen using highly active antiretroviral therapy (HAART) to maximally suppress maternal viral load in the late antenatal period and during the first six months of lactation is safe, effective and can be implemented in resource poor settings in order to reduce the risk of HIV transmission to the infant.

Study Design: The study will be an open label Phase II trial of Zidovudine/Lamivudine and depending on maternal CD4 count, either Nevirapine or Nelfinavir to assess the safety, tolerance and activity of maternal HAART to reduce the risk of transmission among breastfeeding HIV infected women in Kisumu Kenya.

Justification: Transmission through breastfeeding accounts for 25-40% of all mother-to-child transmission of HIV. This trial will assess the safety and activity of a potent triple drug combination to lower maternal viral loadprenatally, intrapartum and during breast feeding. The regimen will be given to HIV infected women from 34 weeks gestation through 6 months of breastfeeding postpartum. Infants will receive a single dose of NVP. Women will be encouraged to breastfeed exclusively and wean abruptly at 6 months. Mother and infant will be followed for 24 months. Clinical and laboratory evaluations will be performed periodically to determine infection status of the infant and side effects of medications to mother and infant. The estimated sample size needed to address both transmission reduction of HAART in comparison to single dose NVP as well as related safety of the two HAART regimens is 520 mother-infant pairs. Comparison will be made with data from previous studies (HIVNET O12 in Uganda and the malaria vertical transmission study in Kisumu) and with data from current Prevention of Mother to Child Transmission (PMCT) programs in Kisumu.

Expectations and significance: A HAART regimen of this nature may potentially show a dramatic decrease in transmission when compared to existing PMCT regimens. Given the continued decreasing costs of ARVs and the relatively low efficacy of existing PMCT regimens, such a regimen would be seriously considered for wide implementation in resource poor settings and elsewhere.

ELIGIBILITY:
Inclusion Criteria:

1. Be a pregnant HIV-infected female presenting prior to 34 weeks gestation who has already chosen to breastfeed after receiving counseling on infant feeding choices according to UNAIDS guidelines which includes counseling and education about the overall benefits of breast feeding as well as the risks of HIV transmission to the infant inherent in breastfeeding.
2. Report that they plan to reside in Kisumu for the next 2 years
3. Be able to give competent, informed consent if >18 or have a parent or guardian who can do the same in the case of a minor.
4. Be willing to comply with study requirements if they meet study eligibility criteria.
5. Meet the following laboratory criteria at enrollment (Efforts will be made to address potentially correctable abnormalities such as anemia, prior to enrollment)

   1. Documentation of HIV-1 infection according to the Kenyan National PMCT testing algorithm.
   2. Serum creatinine <1.5 mg/dl
   3. Hgb >7.0 g/dL
   4. Absolute neutrophil count > 1000 cells/ml
   5. Platelet count >50,000/ml
   6. SGPT < 2.5 times upper limit of normal
   7. Documentation of CD4 count results prior to beginning study drug; which will be used to determine the appropriate HAART regimen -i.e ZDV/3TC/NVP or ZDV/3TC/NLF
   8. Documentation of Hepatitis B and C infection status (Hepatitis B surface antigen and Hepatitis C antibody)
6. Have signed consent and met clinical and laboratory eligibility criteria in order to be enrolled in the trial by 34-36 weeks gestation (preferably at 34 weeks).

Exclusion Criteria:

1. Is participating in other HIV vaccine or antiretroviral trials.
2. Has substantial hypersensitivity to any benzodiazepine, including Nevirapine.
3. Has history of prior substantial intolerance or severe allergic reaction to Nevirapine, Zidovudine, Lamivudine or Nelfinavir.
4. For women who will be placed on NVP, ongoing treatment with rifampin, anticoagulants, benzodiazepines, and magnesium sulfate at time of planned enrollment. For those women who will be placed on NLF, ongoing treatment with amiodarone, quinidine, ergot derivative drugs, rifampin, pimozide, St John's work, lovastatin, simvastatin, midazolam or triazolam
5. Has evidence of clinically significant cardiac, respiratory, hepatic, gastrointestinal, endocrine, hematologic, psychiatric, neurologic, or allergic disease that would compromise the ability of the participant to complete the study or the study requirements as determined by the principal investigator or designated associate. The clinical significance of any abnormality is to be evaluated in the context of the safety of the patient volunteer and the objectives of this study.
6. Has a history of cytotoxic chemotherapy within one month prior to study entry or current diagnosis of malignancy for which systemic therapy is expected to be required during the period of study.
7. Blood pressure > 160 mm Hg systolic or > 110 mm Hg diastolic.
8. Chronic alcohol or illicit drug use.
9. Women who become pregnant again during the study follow-up will NOT be eligible for re-enrollment in the trial if they were enrolled for their previous pregnancy.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2003-07; Primary Completion 2009-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
1. To estimate the cumulative risk of infant infection at 6 weeks, 9 months, and 18 months of age among breast fed infants. The anticipated outcome is a transmission rate of <6% at 6 weeks and <8% at 18 months of age. | 6 weeks, 9 months, 18 months

SECONDARY OUTCOMES:
1. To determine infant HIV-free survival rates at 24 months of age. | 24 months
2. To evaluate infant and maternal safety, and tolerance of ZDV/3TC and Nevirapine or Nelfinavir given to HIV-infected pregnant women from 34 weeks gestation to 6 months postpartum | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy K Thomas, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- CDC Clincical Research Center, Kisumu, Kenya

REFERENCES:
- [Derived] Zeh C, Weidle PJ, Nafisa L, Lwamba HM, Okonji J, Anyango E, Bondo P, Masaba R, Fowler MG, Nkengasong JN, Thigpen MC, Thomas T. HIV-1 drug resistance emergence among breastfeeding infants born to HIV-infected mothers during a single-arm trial of triple-antiretroviral prophylaxis for prevention of mother-to-child transmission: a secondary analysis. PLoS Med. 2011 Mar;8(3):e1000430. doi: 10.1371/journal.pmed.1000430. Epub 2011 Mar 29. PMID 21468304
- [Derived] Thomas TK, Masaba R, Borkowf CB, Ndivo R, Zeh C, Misore A, Otieno J, Jamieson D, Thigpen MC, Bulterys M, Slutsker L, De Cock KM, Amornkul PN, Greenberg AE, Fowler MG; KiBS Study Team. Triple-antiretroviral prophylaxis to prevent mother-to-child HIV transmission through breastfeeding--the Kisumu Breastfeeding Study, Kenya: a clinical trial. PLoS Med. 2011 Mar;8(3):e1001015. doi: 10.1371/journal.pmed.1001015. Epub 2011 Mar 29. PMID 21468300
- [Derived] Harris JR, Greene SK, Thomas TK, Ndivo R, Okanda J, Masaba R, Nyangau I, Thigpen MC, Hoekstra RM, Quick RE. Effect of a point-of-use water treatment and safe water storage intervention on diarrhea in infants of HIV-infected mothers. J Infect Dis. 2009 Oct 15;200(8):1186-93. doi: 10.1086/605841. PMID 19758095